CLINICAL TRIAL: NCT02166164
Title: Characterization of Secondary Hyperalgesia in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Sejer Hansen, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SM1-MSH-2014
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Experimental Pain in Healthy Males
Keywords: Pain; Secondary hyperalgesia; thermal sensitization; Catastrophization; Anxiety
MeSH Terms: conditions — Pain; Hyperalgesia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experiemental pain models (Experimental): all study participants will be tested with the same experimental pain models: Brief thermal sensitization, Long thermal stimulation, and Heat-pain-detection threshold.
  Interventions: Other: Brief thermal sensitization; Other: Long thermal stimulation; Other: Heat-pain-detection threshold

INTERVENTIONS:
Other: Brief thermal sensitization — A small area of the skin of the study participants are heated to 45 degree celsius for 3 minutes, followed by evaluation of secondary hyperalgesia.
  Other Names: Experimental thermal pain model
Other: Long thermal stimulation — A small area of the skin of the study participants are heated to 45 degrees celsius for 1 minute. During the 1 minute period, the study participant will continually report pain on an electronic visual analog scale.
  Other Names: Experimental pain model
Other: Heat-pain-detection threshold — The threshold for heat pain are evaluated by heating a small area of the study participants skin. When the study participant feels pain, the temperature (degrees celsius) is registered.
  4 threshold measurements per session. Heat pain threshold is defined as the average temperature of the 4 measurements.
  Other Names: Experimental pain model

SUMMARY:
In this prospective trial we aim to investigate the intra-individual and inter-individual variance in secondary hyperalgesia following pain elicited by the experimental pain model: Brief Thermal Sensitization.

Furthermore we wish to investigate how precise the psychological tests, Pain Catastrophizing Scale and Hospital Anxiety and Depression Scale predict the size of the area of secondary hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <35 years
* Speak and understand Danish
* Male gender
* Test subjects who have understood and signed the informed consent
* No prescription medicine during the last 30 days

Exclusion Criteria:

* Test subjects that cannot cooperate to the test
* Test subjects with an alcohol and/or substance abuse, assessed by the investigator
* Test subjects, who have consumed one or several types of analgesics 2 <days before the study
* Test subjects, who have consumed antidepressant medication during the last 30 days before the study
* Test subjects with chronic pain
* Test subjects with psychiatric diagnoses
* Test subjects with tattoos on the extremities
* Body Mass Index of >30 or <18

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in area of secondary hyperalgesia following brief thermal sensitization | Study day 1, 2, 3, and 4. A minimum of 4 weeks.
  To determine the intra- and inter-individual variance, and the inter- and intra-observer variance of the secondary hyperalgesia areas following brief thermal sensitization on 4 separate experimental days with two different observers.

SECONDARY OUTCOMES:
Score of Pain Catastrophizing Scale | 7 days
  How precise does the score of the Pain Catastrophizing Scale predict the size of the area of secondary hyperalgesia?
Score of Hospital Anxiety and Depression Scale | 7 days
  How precise does the score of the Hospital Anxiety and Depression Scale predict the size of the area of secondary hyperalgesia?
Score of Subscales of Pain Catastrophizing Scale and Hospital Anxiety and Depression Scale | 7 days
  How precise do the subscales in the two psychological tests (PCS-rumination, PCS-magnification, PCS-helplessness, and HADS-Anxiety, HADS-Depression) predict the size of the area of secondary hyperalgesia?
Heat-pain-detection threshold registered by degrees celsius | 1 minute per session
  How precise do the Heat-pain-detection threshold evaluated on the 4 experimental days predict the size of the area of secondary hyperalgesia on the respective 4 experimental days? 4 sessions of Heat-pain-detection threshold on 4 separate experimental days with 1 session per experimental day.
Pain following Long Thermal Stimulation, evaluated by maximum on the visual analog scale | 1 minute per session
  How precise does the Max. VAS-score following Long Thermal Stimulation evaluated on the 4 experimental days predict the size of the area of secondary hyperalgesia on the respective 4 experimental days? 4 sessions of Long Thermal Stimulation on 4 separate experimental days with 1 session per experimental day.
Pain following Long Thermal Stimulation, evaluated by Area under the curve of the visual analog scale. | 1 minute per session
  How precise does the VAS-Area Under the Curve following Long Thermal Stimulation evaluated on the 4 experimental days predict the size of the area of secondary hyperalgesia on the respective 4 experimental days? 4 sessions of Long Thermal Stimulation on 4 separate experimental days with 1 session per study day.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B Dahl, MD, Doc. Med, Consultant, Study Director — Department of anaesthesiology, dep. Z, Bispebjerg Hospital, Denmark
Locations (1):
- Department of anaesthesia and surgery, 4231, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen MS, Wetterslev J, Pipper CB, Ostervig R, Asghar MS, Dahl JB. The Area of Secondary Hyperalgesia following Heat Stimulation in Healthy Male Volunteers: Inter- and Intra-Individual Variance and Reproducibility. PLoS One. 2016 May 11;11(5):e0155284. doi: 10.1371/journal.pone.0155284. eCollection 2016. PMID 27167119